CLINICAL TRIAL: NCT02256930
Title: A Phase 1, Randomized, Evaluator Blinded, Controlled Study to Evaluate the Sensitizing Potential of M518101 in Healthy Volunteers Using a Repeat Insult Patch Test Design
Brief Title: Skin Safety Study to Evaluate the Sensitizing Potential in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho North America Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: M518101-US07
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sodium Dodecyl Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- M518101 (Experimental): M518101 will be applied 9 times for 21 days on the infrascapular area of the back under occlusive patch conditions.
  Interventions: Drug: M518101
- M518101 Vehicle (Placebo Comparator): M518101 Vehicle will be applied 9 times for 21 days on the infrascapular area of the back under occlusive patch conditions.
  Interventions: Drug: M518101 Vehicle
- Sodium lauryl sulfate (Active Comparator): The sodium lauryl sulfate will be applied 9 times for 21 days on the infrascapular area of the back under occlusive patch conditions.
  Interventions: Other: Sodium lauryl sulfate
- Saline (Sham Comparator): The saline will be applied 9 times for 21 days on the infrascapular area of the back under occlusive patch conditions.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: M518101
  Arms: M518101
Drug: M518101 Vehicle
  Arms: M518101 Vehicle
Other: Sodium lauryl sulfate
  Arms: Sodium lauryl sulfate
Other: Saline
  Arms: Saline

SUMMARY:
This is a single center, randomized, controlled, within subject comparison, multiple dose study to determine the sensitization potential of M518101 on normal skin under occlusive patch condition.

DETAILED DESCRIPTION:
During the Induction Phase of the study, the study drugs and controls will be applied 9 times for 21 days on the infrascapular area of the back under occlusive patch conditions.

Following induction, subjects will have a 10 to 14-day Rest phase, after which they will enter the challenge Phase, which consists of one 48-hour patch application (occlusive) to a naïve site on the opposite side of the back.

ELIGIBILITY:
Inclusion Criteria:

* Health male or female subjects are age 18 years or older
* Signed and dated Informed Consent Form obtained prior to any study related activities
* Subjects are free of any systemic or dermatologic disorder
* For female, females of non childbearing potential or who agree to use a highly effective method of birth control during the study and have a negative urine pregnancy test
* Subjects must be able to communicate with the investigator and understand and comply with the requirement of the study and visit schedule

Exclusion Criteria:

* Have any visible skin disease at the application site which will interfere with the evaluation of the test site reaction
* Have damaged skin in or around the test sites
* Have a history of sensitivity to adhesive tape
* Have a known sensitivity to constituents present in the material being evaluated
* Have a history of, or are currently being treated for skin cancer
* Have used any study drug and/or participate in any clinical study within 60 days prior to randomization
* To engage in any type of strenuous exercise
* Are pregnant, breastfeeding, or of childbearing potential and who wish to become pregnant during the study
* Are deemed to be ineligible by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
inflammatory skin response score | 21 days
  Drug application site will be evaluated for sign of inflammatory skin response (e.g. erythema, edema, papules)

CONTACTS AND LOCATIONS:
Locations (1):
- TKL research, Fair Lawn, New Jersey, United States